CLINICAL TRIAL: NCT04884126
Title: Accuracy, Fitness, Compatibility, and Clinical Outcomes of Customized Implants and Prosthesis in Oral and Maxillofacial Reconstruction
Brief Title: Customized Oral and Maxillofacial Reconstruction
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Hongyang Ma, PhD researcher,, KU Leuven
Other Study IDs: S63615
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Prosthesis Failure, Dental; Dental Implant Failed
Keywords: Dental Implants; Mandibular Reconstruction; Mouth Rehabilitation
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- One stage dental implants placement
  Interventions: Procedure: dental implant placement
- Second stage dental implants placement
  Interventions: Procedure: dental implant placement

INTERVENTIONS:
Procedure: dental implant placement — The time of dental implant surgery

SUMMARY:
Regional oral and maxillofacial defects secondary to ablative tissue resection can contribute to severe aesthetic and functional loss, which influences patients' regular life and may cause psychological problems. Microvascular free flaps are considered the gold standard for reconstructing large oral and maxillofacial defects. In the past decade, with the help of computer-aided design (CAD)/ computer-aided manufacturing (CAM) customized implants and prosthesis (CIP) have led to a significant improvement of the operative accuracy, improve the flap survival rate and enhance the patients' quality of life.

Concerning the increased overall survival rate of the patients, people pay more attention to the quality of life and aesthetic appearance which are influenced by the fitness and compatibility of the CIP. However, from literature reviews, the evaluation was various to be concluded in some certain conditions from pooled studies.

DETAILED DESCRIPTION:
The trial will be conducted in compliance with the principles of the Declaration of Helsinki (specifying which amendment), the principles of GCP, and all of the applicable regulatory requirements. This protocol and related documents will the for review to the Ethics Committee. The Investigator and the Participating Site shall treat all information and data relating to the Study disclosed to Participating Site and/or Investigator in this Study as confidential and shall not disclose such information to any third parties or use such information for any purpose other than the performance of the Study. The collection, processing, and disclosure of personal data, such as patient health and medical information is subject to compliance with applicable personal data protection and the processing of personal data (Directive 95/46/EC and Belgian law of December 8, 1992, on the Protection of the Privacy in relation to the Processing of Personal Data). The extracted data will be encoded, the subject's EAD-number will be stored separately(site file) from the research data and replaced with a unique study ID-code to create a new identity for the subject. The file containing the patient-specific EAD-numbers will be kept on a secured UZ Leuven servers.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with grafted bone (fibula, iliac, scapula) and receive postoperative implant surgery.

  2.Clinical and radiogram data were available for all treatment periods and follow-up visits (Pre-/post-CBCT and panoramic radiographs).

  3.Over twelve months follow-up period after implant placement. 4.Age > 18 years. 5.Fabrication and delivery of prosthesis following implant installation. 6.Treatment with a one-stage/two-stage surgical protocol.

Exclusion Criteria:

1. Patients diagnosed with osteoporosis.
2. Lost or missing medical history during follow-up period.
3. Follow-up period of dental implants was less than 12 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The files of patients diagnosed and treated between December 2004 and January 2020 for defect of dentition secondary to jaw resection were retrospectively reviewed. The patients who underwent dental implant surgery after ablative tumor resection with segmental mandibulectomy and vascularized bone flap graft were retrieved from the database.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 1996-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
The survival rate of the dental implants | 12 months after surgery

IPD SHARING:
Plan to Share IPD: Undecided